CLINICAL TRIAL: NCT01559376
Title: Long Term Follow-up of Open Versus Endoscopic Radial Artery Harvest With CT Angiography
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: ENDO2012
Record Dates: First submitted 2012-02-27; First posted 2012-03-21 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2012-03

CONDITIONS: Arteriosclerosis of Arterial Coronary Artery Bypass Graft

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Endoscopic radial artery harvest
- Conventional open radial artery harvest

SUMMARY:
The objectives of the study are two-fold:

1. To determine the mean 5 year patency rate of the radial artery graft (Open vs. Endoscopic) of patients who have already had CABG surgery and who previously participated in the centre's RCT back in 2005-2007 using CTA and MPS-MIBI
2. To determine patient quality of life at 5 years post CABG surgery

It is hypothesized that the mean 5 year patency rate of the radial artery graft harvested endoscopically will be equal to or have greater patency than the radial artery graft harvested via the conventional/open technique. It is further hypothesized that patient quality of life will be similar amongst patients having had the open vs. endoscopic radial artery graft during CABG surgery.

DETAILED DESCRIPTION:
After patient consent and REB approval from The University of Western Ontario (REB # 11054) we conducted a Randomized Controlled Trial between 2005-2007 of endoscopic vs. conventional harvesting of the radial artery in CABG patients at the London Health Sciences Centre. A total of 118 patients were randomized to either A) conventional/open harvesting of the radial artery, n=59 or B) endoscopic harvesting of the radial artery, n=59. Post-operative study objectives measured were arm wound infection rate, assessment of arm pain, arm edema, mobilization, patient satisfaction, and histological assessment of the radial artery. Objectives were measured during the patients' course in-hospital and at 1week by telephone interview. At 6 weeks patient underwent a final clinic assessment post-surgery.

Our intent is to perform follow-up angiography and MPS-MIBI at the 5 year mark post surgery on the 118 patients previously involved in our RCT, to assess open vs. endoscopic radial artery graft performance. The study will be divided into three phases: Phase I - Patient Recruitment (4 months), Phase II - Patient Assessment with CTA, MPS-MIBI and Questionnaires (16 months) and Phase III - Data Analysis and Conclusions (4 months).

Phase I - Chart Review and Patient Recruitment (4 Months) Charts will be reviewed on all of the open and endoscopically harvested radial artery grafts used during CABG surgery from the above specified time points. Patient demographics and operative notes, as well as perioperative and postoperative complications will be reviewed. Hospital admissions, documented cardiac events and any subsequent deaths not previously documented will be recorded. Any additional pertinent data from the chart review will be entered into a study specific Microsoft Excel file maintained by a single qualified research assistant.

All living CABG surgery patients will then be contacted and their participation in the study requested. Patients will receive an initial request by mail, with an informative letter signed by the principal investigator outlining the purpose of the study, what participation in the study involves, and the specific aims of the cardiac team at the conclusion of the study. A follow-up phone call will be done within 3-weeks of mailing the letter to go over the content and answer any questions that patients may have.

Phase II - Patient Assessment via CTA, MPS-MIBI and Questionnaires (16 Months)

CABG surgery patients from the previous RCT that agree to be a part of the study will have arrangements made for them to travel to LHSC. Patients will undergo a structured half-day (approximately 4-6 hours) at the hospital consisting of the following:

1. Selective coronary artery and radial artery graft check via CTA with a 64 slice CT scanner + Rest MPS-MIBI then Stress MPS-MIBI (4-6hrs). The CT scanner along with the stress/rest MIBI machine are dedicated "Research only" machines. As such, there are no issues with using these research dedicated machines and there is no additional cost to OHIP.
2. Completion of two validated health related quality of life questionnaires

   1. Seattle Angina Questionnaire
   2. 36-Item Short Form Health Survey SELECTIVE CORONARY ARTERY & RADIAL ARTERY GRAFT CHECK VIA CTA AND REST & STRESS MPS-MIBI

Coronary CTA and Rest and Stress MPS-MIBI will be used for evaluating radial artery graft patency. Potential risks associated with CTA and both MPS-MIBI tests will be discussed with each patient prior to performing the procedure. This discussion will include the following:

As CTA is an x-ray test, it sends radiation through the body. Although the amount of radiation for each scan is small, it can accumulate and damage body cells over time with repeated exposure. Contrast material carries a slight risk of causing an allergic reaction to the contrast material or dye. During the Rest and Stress MPS-MIBI, a radioactive tracer (MIBI) is used to take pictures of the heart. This tracer is injected into the bloodstream and travels to the heart muscle through the coronary arteries. Pictures are then taken of the heart to determine coronary artery disease and the perfusion images at rest and stress help identify regions of myocardial infarction as well as help determine the hemodynamic significance of any coronary stenoses. MPS also gives an estimate of the left ventricular ejection fraction. Signed consent will be obtained prior to each procedure. Contrast will be injected into the coronary arteries and the vein grafts and CTA and MPS-MIBI images obtained.

EVALUATING RADIAL ARTERY GRAFT PATENCY All coronary artery and radial artery graft CTAs and MPS-MIBIs will be performed and graded by Nuclear Medicine physicians. Following the patency determination, the patients will be contacted by Dr.Bob Kiaii (cardiac surgeon) and told their results.

Radial artery graft patency will be determined using the grading system of Fitzgibbons and associates:

Grade A Excellent graft with unimpaired run-off, patent graft Grade B Stenosis reducing caliber of proximal, distal anastomosis or trunk to <50% of the grafted coronary artery. This will be divided into flow limiting and non-flow limiting stenosis Grade O Occlusion

QUALITY OF LIFE QUESTIONNAIRES To assess quality of life 5 years after undergoing CABG surgery and participating in our RCT, each patient will self-administer two validated health-related quality of life questionnaires while on site at LHSC. The two questionnaires to be used are the Seattle Angina Questionnaire (SAQ) and the 36-Item Short Form Health Survey. Licensing and user registration permitting use of these questionnaires will be obtained online from Cardiovascular Outcomes Inc. (SAQ) and Quality Metric (SF-36) prior to their distribution and use.

SEATTLE ANGINA QUESTIONNAIRE The SAQ is a 19-item, well standardized self-administered questionnaire shown to be a valid measure of quality of life in patients suffering from coronary artery disease. The disease-specific questionnaire measures five clinically important dimensions of health in coronary artery disease patients: physical limitations, angina stability, angina frequency, treatment satisfaction and disease perception. The SAQ has shown to be more sensitive to clinical change in coronary artery disease in comparison to more generic quality of life questionnaires.

36-ITEM SHORT FORM HEALTH SURVEY The SF-36 is a 36-item, generic quality of life questionnaire for measuring patient's general health status. Also well-standardized and self-administered, the SF-36 measures eight health concepts: physical conditioning, role limitations due to physical problems, social functioning, bodily pain, and general mental health, role limitations due to emotional problems, vitality and general health perceptions. It also includes an indication of perceived change in health. The questionnaire has proven relevant across age, disease process and treatment group.

Using a disease-specific questionnaire and a general health questionnaire in combination will more aptly categorize the overall impact of the CABG surgery on patient quality of life. The effects of CABG surgery both in regards to cardiovascular function as well as outside systems will be better understood.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they:

  1. Have previously participated in our RCT from 2005-2007 with an open or endoscopically harvested radial artery graft used as a bypass conduit.
  2. Willing to give informed consent to participate in the study

Exclusion Criteria:

* Patients are excluded if they are:

  1. Expired
  2. Unable or unwilling to give informed consent
  3. History of allergic reaction to contrast material used in CTA or severe adverse reactions to medications used in MPS-MIBI procedures
  4. Kidney dysfunction

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The patient population consists of patients that have previously participated in our RCT from 2005-2007 with an open or endoscopically harvested radial artery graft used as a bypass conduit. We are following them for 5-year follow up.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Radial artery graft patency | Mean 5 years
  Grade A Excellent graft with unimpaired run-off, patent graft Grade B Stenosis reducing caliber of proximal, distal anastomosis or trunk to <50% of the grafted coronary artery. This will be divided into flow limiting and non-flow limiting stenosis Grade O Occlusion

SECONDARY OUTCOMES:
Ischemia present in other coronary artery territories | Mean 5 years
  Areas of decreased perfusion identified by MPS-MIBI scanning in the context of CT - angiographic results
Identification of left ventricular ejection fraction at rest and stress | Mean 5 years
  Related in percentage of blood ejected as a fraction of left ventricular end diastolic volume
Quality of life post CABG via the two questionnaires; the Seattle Angina Questionnaire (SAQ) and the 36-Item Short Form Health Survey. | Mean 5 years
  Numerical score based on the questionnaire scoring scales
Stenosis present in other coronary arteries / grafts | Mean 5 year
  Based on CT - angiographic results. Grade A: unimpaired run-off, patent graft Grade B Stenosis reducing caliber of proximal, distal anastomosis or trunk to <50% of the grafted coronary artery. This will be divided into flow limiting and non-flow limiting stenosis Grade O Occlusion

CONTACTS AND LOCATIONS:
Overall Officials: Bob Kiaii, BSc, MD, Principal Investigator — University of Western Ontario, Lawson Research Institute, University of Western Ontario
Locations (2):
- Canada (2):
  - London Health Sciences Centre, University Hospital, London, Ontario
  - London Health Sciences Centre, Victoria Hospital, London, Ontario